CLINICAL TRIAL: NCT05541666
Title: Effect of Emotional Freedom Technique on Postoperative Pain and Anxiety in Patients Undergoing Total Knee Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Pınar Tanrıver, Research assistant, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ATAUNIYLTEZTANRIVER-001
Record Dates: First submitted 2022-09-13; First posted 2022-09-15 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Total Knee Arthroplasty
Keywords: Anxiety; Emotional Freedom Technique; Pain; Total Knee Replacement
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Intervention Model Description: This study was planned as a parallel, two-arm randomized controlled trial (RCT).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): EFT will applied to the patients in the experimental group on the 1st and 2nd days after surgery.
  Interventions: Other: Emotional Freedom Technique (EFT)
- Control Group (No Intervention): Patients in the control group will received no treatment other than the clinic's routine patient care.

INTERVENTIONS:
Other: Emotional Freedom Technique (EFT) — EFT is an energy psychology intervention that utilizes cognitive behavioral therapy, exposure therapy, and acupuncture points to create psychological and physical changes in individuals. It is also referred to as "acupuncture without needles" or an emotional form of acupressure.
  Arms: Experimental group

SUMMARY:
The purpose of the present study was to examine the effects of the Emotional Freedom Technique on pain and anxiety in the postoperative period of patients who underwent total knee arthroplasty.

Research Hypotheses H1: Emotional freedom technique reduces postoperative pain level in patients undergoing total knee arthroplasty.

H2: Emotional freedom technique reduces postoperative anxiety level in patients undergoing total knee arthroplasty.

DETAILED DESCRIPTION:
One day before the surgery the patients in both groups will interviewed and the Patient Descriptive Data Form, Visual Analog Scale (VAS) Pain, and State Anxiety Inventory (SAI) will applied. Then, information will given to the experimental group about EFT and the patients' questions will answered. On the first postoperative day between 18.00 and 20.00 the patients in both groups will interviewed to collect the pretest data and VAS Pain, SAI, and Subjective Unit of Experience Scale (SUE) will applied. Then, the EFT steps will explained and demonstrated to the experimental group and a session of EFT will applied. After the EFT, the SUE Scale will re-evaluated without any break. On the second postoperative day between 18.00 and 20.00 the patients in both groups will interviewed again, and the SUE Scale will evaluated. Then, a session of the EFT will applied to the experimental group. After the EFT, VAS Pain, SAI, and SUE will re-applied without any break for post-test data. In the control group VAS Pain, SAI, and SUE will re-applied for post-test data on the second postoperative day between 18.00 and 20.00.

ELIGIBILITY:
Inclusion Criteria:

1. Elective patients undergoing total knee replacement surgery for the first time,
2. Volunteer to participate in the research,
3. 18 years and over,
4. Cognitive level scales are suitable for application,
5. Having no vision, hearing, or speech problems that would prevent communication,
6. Patients who do not have any other disease causing pain and anxiety

Exclusion Criteria:

1. EFT was applied before,
2. If any complication develops within 3 days before, during, or after the operation,
3. Patients with health problems (fever, infection, deep vein thrombosis, etc.) that prevent the application of the Emotional Freedom Technique were not included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-03-07 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2023-01-02 (Actual)

PRIMARY OUTCOMES:
anxiety level | Post-operative 1st and 2nd day
  On the postoperative 1st day and 2nd day, patient's anxiety status will evaluated with State Anxiety Inventory (SAI)
pain level | Post-operative 1st and 2nd day
  On the postoperative 1st day and 2nd day, patient's pain status will evaluated with Visual Analog Scale (VAS).

CONTACTS AND LOCATIONS:
Overall Officials: Dilek Gürçayır, Principal Investigator — Ataturk Univesity; Dilek Gürçayır, Principal Investigator — Ataturk University
Locations (1):
- Atatürk University, Erzurum, Yakutiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No